CLINICAL TRIAL: NCT04581057
Title: Frequency of Clonal Hematopoiesis in Patients Over 75 With a First Cardio Vascular Event. Consequences on Inflammation and Atherosclerosis
Brief Title: Correlation Between Clonal Hematopoiesis, Cardio-vascular Events, Inflammation and Atherosclerosis
Acronym: CHATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2019/18
Record Dates: First submitted 2020-10-02; First posted 2020-10-09 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Myocardial Infarction
Keywords: CHIP; Cardiovascular events; Atherosclerosis; Inflammation
MeSH Terms: conditions — Myocardial Infarction; Atherosclerosis; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First CVE (Experimental)
  Interventions: Biological: Specific blood sampling

INTERVENTIONS:
Biological: Specific blood sampling — A 30 ml blood sample (6 EDTA tubes) will be taken at inclusion in the study, in addition to the blood sample taken as part of the routine care.
  This sampling is carried out for :
  * Search for CHIP-associated mutations in circulating leukocytes
  * Plasma determination of IL-1β, IL-6, IL-10 and TNF-α

SUMMARY:
This study aims at evaluating the prevalence of Clonal Hematopoiesis of Indeterminate Potential (CHIP) in patients over 75 presenting with a first cardio-vascular event (CVE). The investigators will also determine if CHIPs are more frequent in this population compared to a control cohort without CVE. An association between CHIP, a systemic inflammation and increased atherosclerosis will also be assessed.

DETAILED DESCRIPTION:
Despite increasing knowledge on the pathophysiology of cardio-vascular diseases (in particular the role of inflammation in the development of atherosclerosis), predicting their occurrence remains largely difficult. Aging remains the most powerful factor for predicting the occurrence of myocardial infarction, independently from other identified risk factors. Few years ago, acquired mutations were described in the hematopoietic system of apparently healthy subjects. This phenomenon, now described as CHIP (Clonal Hematopoiesis of Indeterminate Potential) is more frequently observed in elderly people, and has been recently linked to an increased risk of cardio-vascular events. Experiments in mice demonstrated that these CHIPs are responsible for an inflammation that supports the development of atherosclerosis. However the link between CHIP, inflammation and atherosclerosis has never been demonstrated in humans.

In this study, the investigators will search for an increased frequency of CHIP in patients with a first cardio-vascular event (CVE). Seven months after the CVE, a blood sample will be taken. Mutations in the 9 most frequently mutated genes in CHIP will be evaluated by Next Generation Sequencing. Systemic inflammation will be evaluated by measurement of circulating levels of CRP, IL-1β, IL-6, IL-10 and TNF-α. Atherosclerosis will be evaluated via the volume of atherosclerotic plaques as assessed by 3D ultrasound analysis. The presence of CHIP will be correlated to traditional cardiovascular risk factors, systemic inflammation markers and the level of atherosclerosis. The investigators will also assess the relationship between the presence of CHIP and the risk of CVE reoccurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) over 75 years old
* Patients with a first CVE (myocardial infarction) of atheromatous origin that occurred between 2 and 7 months before inclusion
* Absence of evidence of hematological malignancy (known or obvious by the results of blood counts)
* Subject registered with a social security scheme
* Written informed consent obtained

Exclusion Criteria:

* Patients who did not presented any CVE in the last 7 months
* Patients with CVE with a non-atheromatous origin (dissection, embolic, …)
* Presence of an unbalanced diabetes (defined as HbA1C > 10%)
* History of previous CVE before 75 year-old : myocardial infarction, stroke of atheromatous origin
* Hematological malignancy (known or obvious on the results of blood counts)
* Chronic inflammatory disease (cancer, vasculitis, rheumatism, hepato-gastro-intestinal diseases).
* Long term anti-inflammatory treatments:

  * Corticoids
  * Nonsteroidal anti-inflammatory drugs
  * Aspirin (> 325 mg per day)
  * Cyclo-oxygenase II inhibitors
* Persons under judicial safeguards, trustee or curators
* Person deprived of judicial or administrative freedom
* Person unable to give her consent
* Non-cooperative person
* Exclusion period after another clinical study or participation to another interventional clinical study testing a drug in the 30 days before inclusion

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-10-03 (Actual); Study Completion 2021-10-03 (Actual)

PRIMARY OUTCOMES:
Presence of a CHIP | Day 1
  Defined as the presence of a mutation (in the genes DNMT3A, TET2, ASXL1, SF3B1, TP53, CBL, SRSF2, GNB1 and PPM1D) (with an allelic frequency greater than 2, 5 or 10%).

SECONDARY OUTCOMES:
Frequency of CHIP | Day 1
  The frequency of CHIP in this cohort will be compared to the one observed in a control population (recruited from the 3-cities study cohort or 3C).
Assessment of systemic inflammation | Day 1
  Assessed by the level of plasmatic CRP, IL-1β, IL-6, IL-10 and TNF-α.
Assessment of Atherosclerosis level | Day 1
  Assessed by 3D ultrasound analysis. An innovative technique for monitoring the volume of carotid plaques.
Presence of cardiovascular risk factor | Day 1
  Evaluated by the investigators.The cardiovascular risk factor are defined as :
  * Active smoking or smoking cessation for less than 3 years
  * HyperLDLemia (LDL Cholesterol > 3.36 mmol/L)
  * HypoHDLemia (HDL < 1.03 mmol/L in men or < 1.29 mmol/L in women)
  * Diabetes (2 blood glucose levels > 6.93 mmol/L)
  * Hypertension (hypertension) (> 140/90 mmHg) treated or not.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry COUFFINHAL, MD-PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fawaz S, Marti S, Dufossee M, Pucheu Y, Gaufroy A, Broitman J, Bidet A, Soumare A, Munsch G, Tzourio C, Debette S, Tregouet DA, James C, Mansier O, Couffinhal T. Evaluation of clonal hematopoiesis and mosaic loss of Y chromosome in cardiovascular risk: An analysis in prospective studies. Elife. 2024 Dec 12;13:RP96150. doi: 10.7554/eLife.96150. PMID 39665621